CLINICAL TRIAL: NCT01943630
Title: A Phase II, Multicenter, Randomized, Double Blind, Vehicle Controlled Study Evaluating the Efficacy and Tolerability of AS101 15% Gel for External Genital Warts.
Brief Title: Safety and Efficacy Double Blind Vehicle Controlled Study of 15% AS101 Gel to Treat External Genital Warts
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioMAS Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS101-IL#002
Record Dates: First submitted 2013-09-09; First posted 2013-09-17 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: External Genital Warts
Keywords: HPV condyloma acuminata

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AS101 (Active Comparator): Topical 15% AS101 gel, once a day (overnight)
  Interventions: Drug: 15% AS101 gel
- Vehicle (Placebo Comparator): Vehicle, Once a day topical application (Overnight)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: 15% AS101 gel — Administration of Topical 15% AS101 once a day (overnight)
  Arms: AS101
Drug: Vehicle — Administration of Vehicle once a day (overnight)
  Arms: Vehicle

SUMMARY:
The purpose of this double blind study is to determine whether topical 15% AS101 gel is effective and safe as compared to vehicle in the treatment of external genital warts in women.

DETAILED DESCRIPTION:
Females with external genital warts who meet the eligibility criteria will be randomly allocated in a blinded manner in 1:1 ratio to one of the 2 following study arms: (1) AS101 15% gel or (2) Vehicle. The patients will apply the study drug at home once daily (overnight) until complete clearance of external genital warts or for up to 14 weeks (98 days).

During therapy all patients will return to the clinic every 2 weeks plus/minus 3 days of the treatment visit for clinical assessments of the treated area.

At week 6 of treatment the investigator will evaluate the treated area for all patients. If the investigator determines that there is no change in the disease spread area or lesion number compared to Day 1, study therapy is to be discontinued prior to 14 weeks (98 days) of treatment and the patient will be considered as not cleared. Last observation carried forward (LOCF) method will be used to analyze such patients.

Patients who at week 6 were evaluated by the investigator to have a change in the disease spread area or lesion number compared to Day 1, will continue treatment until complete clearance of warts or up to a maximum of 14 weeks (98 days).

Patients who were evaluated during any of the treatment visits with complete clearance will stop to apply the study therapy, continue to be followed once per 4 weeks for 84 days (12 weeks) for safety and recurrence evaluation. Patients who completed treatment with partial clearance or patients who discontinued for reasons of other than complete clearance will be followed 28 days after discontinuation for disease progression and reference to other therapy if was recommended.

Should significant irritation or any other skin adverse reaction occur during the treatment period, study therapy may be held for up to 7 consecutive days on up to two separate occasions.

Unblinding: Patients will be revealed as to the nature of their treatment only after all patients have completed study.

In case of pregnancy or related serious adverse event the nature of the treatment will be revealed to the patient prior to end of study.

If the investigator determines that there is a disease progression in total lesion number or infected wart area size of the Day 1 treated area, study therapy is to be discontinued prior to 98 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women at least 18 years of age and in good health;
2. Must sign an ethics committee approved informed consent form and be able to adhere to study visits and protocol requirements;
3. Women must agree to avoid sexual contact while the gel is on their skin;
4. All study participants who are sexually active must use a protection method of contraception during treatment and for 60 days after completion of treatment;
5. Patients with clinical diagnosis of external genital warts, in the external genitalia including vulva (labia minora and majora), inguinal folds, pubic area, perineum, perianal, or buttocks areas; two or more distinct external genital warts, and wart area to be treated that is equal to or less than 10 cm2.

Exclusion criteria:

1. Participation in an investigational trial within 30 days prior to screening;
2. Previous participation in a trial investigating AS101 for any indication;
3. Topical treatment for genital warts within 14 days of screening;
4. Cutaneous surgery, including cryosurgery or laser, to genital area within 30 days of screening;
5. Skin irritations of other clinical signs or symptoms associated with prior therapy.
6. Topical and systemic immunosuppressive or immunomodulatory medications (including corticosteroids) within 30 days prior to screening, and while on study;
7. Current active infection with herpes genitalis or history of herpes genitalis infection within the last 30 days prior to screening (patients on long-term suppressive antiviral therapy are eligible);
8. Diagnosis of high-grade cervical dysplasia;
9. Internal anogenital, vaginal, cervical warts or urethral meatal warts requiring treatment;
10. Chronic or acute skin condition that might interfere with the treatment or evaluation of study drug effect;
11. Screening laboratory tests results from a complete blood count (CBC), chemistry panel and urine pregnancy test obtained during screening:

    1. Must be within the site laboratory's defined normal reference ranges, and/or according to the Investigator's decision;
    2. Urine pregnancy test in females of childbearing potential must be negative;
    3. Inadequate renal function: Serum Creatinine >2.0mg/dL (>2.0 ULN);
    4. Inadequate liver function: Serum (total) Bilirubin >2 mg/dl or ALT and/or AST greater than two times the upper limit of the reference range.
12. Uncontrolled infection or acute severe febrile illness;
13. Diagnosed as having uncontrolled cardiovascular, hematological, hepatic, neurological, renal, endocrine, vascular, autoimmune, or gastrointestinal abnormalities or disease;
14. Pregnant or lactating;
15. Known allergy to AS101 or any component of the investigational formulation; or
16. Subjects with any other clinically significant medical condition, psychiatric condition or laboratory abnormality which would, in the judgment of the Investigator, interfere with the subject's ability to participate and comply with the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in number of warts and infected area size (absolute and percent) as compared to Day 1. | within 14 weeks of treatment

SECONDARY OUTCOMES:
Assessment of safety of AS101 15% gel as expressed by the occurence of local topical reactions such as erythema and edema and systemic reactions to the treatment | within 14 weeks of treatment and 3 months of follow up
In complete responders assessment of time to complete clearance of warts. | within 14 weeks of treatment
In complete responders assessment of recurrence rate and time to recurrence. | Within 3 months of follow up post treatment
Collection of patient's satisfaction data from treatment etc. | within 14 weeks of treatment
Assessment of tolerability to the 15% AS101 gel as expressed by patient's itching and burning reports. | within 14 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shabtai Romano, MD, Principal Investigator — Ha'Emek Medical center, Department of Gynecology & obstetrics
Locations (4):
- Israel (4):
  - Ha'Emek Medical Center, Department of Gynecology and obstetrics, Afula
  - Kaplan Medical Center, Department of Gynecology, Rehovot
  - Ziv Medical Center, Department of Gynecology and obstetrics, Safed
  - Tel-Aviv Sourasky Medical Center, Department of Gynecology, Tel Aviv